CLINICAL TRIAL: NCT00406939
Title: Phase I Study of Adenoviral Vector Delivery of The IL-12 Gene in Men With Recurrence or Persistent Cancer of the Prostate After Primary Therapy With or Without Metastatic Disease (SPORE)
Brief Title: Vector Delivery of the IL-12 Gene in Men With Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Baily, Baylor College of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #H-6836; P50CA058204 (NIH)
Record Dates: First submitted 2006-12-01; First posted 2006-12-04 (Estimated); Last update posted 2008-07-10 (Estimated); Status verified 2008-07

CONDITIONS: Prostatic Neoplasms; Prostate Cancer
Keywords: Gene Therapy; Immunology; Phase I Clinical Trial
MeSH Terms: conditions — Prostatic Neoplasms

INTERVENTIONS:
Genetic: IL-12 gene

SUMMARY:
This study is designed to determine the safety of IL-12 gene therapy for patients with recurrence of prostate cancer after radiation therapy and those with or without metastatic disease with a prostate gland intact. These, of course, would include recurrent prostate cancer after definitive radiation therapy. The prostate cancer will be treated with a prostatic injection of a replication-defective adenovirus vector delivering the IL-12 gene. Following virus injection, patients will be hospitalized for 23 hours for observation. Only one course of therapy will be administered. Each patient will be carefully monitored for toxic effects. Three to five patients will be tested with a low dose of virus and if there are no serious adverse side effects, the dose will be slowly escalated in subsequent groups of 3-5 patients or until unacceptable toxicity is reached. Effectiveness will be monitored by serum prostate-specific antigen (PSA), transrectal ultrasound of the prostate, prostate biopsy and comparison of survival times to historical survival times for patients with radiation recurrent prostate tumors. The primary objective of this initial study is to determine whether the treatment is associated with significant toxicity.

DETAILED DESCRIPTION:
The development of a clinical trial for gene therapy in prostate cancer will be coordinated with our collaborators at Baylor involved in similar studies in order to facilitate the approval process. We have submitted a proposal to the NIH Recombinant DNA Advisory Committee (RAC) committee for accelerated review. A detailed clinical protocol and informed consent for a Phase I clinical trial of gene therapy for prostate cancer has been approved by the Baylor Affiliates Review Board and the FDA.

Human subjects included in this project will be limited to men who have biopsy-proven local recurrence or persistence of cancer in the prostate gland with or without metastatic disease after hormone therapy, cryosurgery and/or definitive irradiation therapy. Patients with biopsy-proven prostate cancer, clinical stages T1-T3, Nx-N1 or M0-M1 are eligible. Biologically active local recurrence of tumor will be defined as biopsy-proven cancer in the prostate, at least one year after the completion of radiation therapy, in a patient who has a rising serum PSA level on at least 3 separate occasions at least 2 weeks apart.

Patients will also be carefully followed to document toxicity, using standard CTEP toxicity criteria. Responses will be categorized as follows: progressive disease, stable disease, partial objective response, and complete objective response. Progressive disease will be defined as a rise in the serum PSA level by 25% in the first 3 months and thereafter, a positive biopsy in conjunction with an enlarging nodule on digital rectal exam or an enlarging hypoechoic lesion on ultrasound, or the development of new symptoms clearly related to the cancer in the presence of a positive biopsy, or the presence on biopsy of cancer of higher grade or cancer that is more extensive. A complete response will be defined as a serum PSA level that decreases to less than 1 ng/ml, in combination with a negative biopsy of the prostate and the absence of symptoms referable to cancer. A partial objective response would be a PSA level that decreases by at least 50% compared to baseline in association with a biopsy result that shows clearly diminished or minimum but persistent cancer cells.

This Phase I study is designed to evaluate the safety of Adv/IL-12 gene therapy with an intent to offer a potential therapeutic advantage. The potential risks associated with the use of gene therapy in this group would appear reasonable in so far as evaluations will be frequent and progression (should it occur) will be found early and allow rapid movement of the patient to other possible therapies. Effectiveness will be monitored by serum PSA, transrectal ultrasound of the prostate, prostate biopsy and comparison of survival times to historical survival times for patients with radiation recurrent prostate tumors. Additional research laboratory analyses will be performed to evaluate the immune response engendered by this gene therapy protocol. This will consist of analysis of serum and/or plasma and urine for systemic cytokine production using standard ELISA methodologies that we have performed in previous studies. In addition we will collect whole blood for the analysis of T cells by flow cytometry. We have established protocols for this analysis that can detect total CD4 and CD8 cells as well as those that express markers of activation such as HLA/DR.

ELIGIBILITY:
Inclusion Criteria:

* Men who have biopsy-proven local recurrence or persistence of cancer in the prostate gland with or without metastatic disease after the hormone therapy, cryosurgery, and/or the completion of definitive radiation therapy for at least one year.
* Patients must have evidence of biologically active local recurrence of tumor as demonstrated by a rising serum PSA level on at least 3 separate occasions at least 2 weeks apart, and that the serum PSA be below 50 ng/ml.
* The patient will possess the ability to give informed consent and express a willingness to meet all the expected requirements of the protocol for the duration of the study. (Informed Consent Document).
* Patients must have adequate baseline organ function as assessed by the following laboratory values before initiating the protocol.

  1. Adequate renal function with serum creatinine less than 1.5 mg/dl or creatinine clearance greater than 45 ml/min/m2.
  2. Platelet count greater than 100,000 platelets/mm3.
  3. Absolute neutrophil count greater than 1000/mm3.
  4. Hemoglobin greater than 8.5 mg/dl
  5. Normal partial thromboplastin time (PTT) and Pro-Thrombin Time (PT).
  6. Bilirubin less than 2.5 mg/dl, SGOT and SGPT less than 2.0x normal.

Exclusion Criteria:

* Acute infection: Acute infection is defined as any viral, bacterial or fungal infection, which requires specific therapy.
* Symptomatic metastasis.
* Metastatic lesions in the CNS/spinal cord or organs that could become life or function threatening within 3 months.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 1998-06; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
To determine whether the treatment is associated with significant toxicity.

SECONDARY OUTCOMES:
Collection of data on tumor responses produced by the study treatment.
Collection data on immune responses induced by the study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Brian J. Miles, M.D., Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine Scott Department of Urology, Houston, Texas, United States

REFERENCES:
- [Background] Shalev M, Kadmon D, Teh BS, Butler EB, Aguilar-Cordova E, Thompson TC, Herman JR, Adler HL, Scardino PT, Miles BJ. Suicide gene therapy toxicity after multiple and repeat injections in patients with localized prostate cancer. J Urol. 2000 Jun;163(6):1747-50. PMID 10799174
- [Background] Fujita T, Timme TL, Tabata K, Naruishi K, Kusaka N, Watanabe M, Abdelfattah E, Zhu JX, Ren C, Ren C, Yang G, Goltsov A, Wang H, Vlachaki MT, Teh BS, Butler EB, Thompson TC. Cooperative effects of adenoviral vector-mediated interleukin 12 gene therapy with radiotherapy in a preclinical model of metastatic prostate cancer. Gene Ther. 2007 Feb;14(3):227-36. doi: 10.1038/sj.gt.3302788. Epub 2006 Oct 5. PMID 17024109
- See also: Scott Department Of Urology Clinical Trials — http://www.baylorurology.org